CLINICAL TRIAL: NCT04052620
Title: A Randomized, Double Blind, Multi Center, Active-controlled, 2 Treatment Arm, Parallel Group Non Inferiority Study to Evaluate the Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel Versus 1.16% Gel in Subjects With Acute Ankle Sprain
Brief Title: Voltaren Emulgel 2% Acute Ankle Sprain Non Inferiority Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 211206; 2016L09875 (Registry Identifier: NMPA)
Record Dates: First submitted 2019-07-23; First posted 2019-08-12 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Pain
Keywords: Ankle sprain; diclofenac diethylamine
MeSH Terms: conditions — Pain; Ankle Injuries | interventions — diclofenac diethylamine; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac diethylamine (DDEA) 2.32%/ Placebo gel (Experimental): Participants will receive 4 tubes, DDEA 2.32% gel and Placebo gel (2 each) and instructed to apply the gel 5 centimeter (cm) topically with the finger tips (for approximately 1 minute) on both sides of affected ankle on area of approximately 200 square centimeters (cm^2). DDEA 2.32% gel will be applied in morning and late afternoon and Placebo gel will be applied in noon and late evening for 7 days.
  Interventions: Drug: Diclofenac diethylamine 2.32% gel; Other: Placebo
- DDEA 1.16% gel (Active Comparator): Participants will receive 4 tubes of DDEA 1.16% gel and instructed to apply the gel 5 centimeter (cm) topically with the finger tips (for approximately 1 minute) on both sides of affected ankle on area of approximately 200 square centimeters (cm^2) in morning, noon, late afternoon, and late evening for 7 days.
  Interventions: Drug: Diclofenac diethylamine 1.16% gel

INTERVENTIONS:
Drug: Diclofenac diethylamine 2.32% gel — Participants will apply DDEA 2.32% gel topically with the finger tips (for approximately 1 minute) on both sides of affected ankle 5 cm on 200 cm^2 two times daily for 7 days.
  Arms: Diclofenac diethylamine (DDEA) 2.32%/ Placebo gel
Drug: Diclofenac diethylamine 1.16% gel — Participants will apply DDEA 1.16 % gel topically with the finger tips (for approximately 1 minute) on both sides of affected ankle 5 cm on 200 cm^2 four times daily for 7 days.
  Arms: DDEA 1.16% gel
Other: Placebo — Participants will apply Placebo gel topically with the finger tips (for approximately 1 minute) on both sides of affected ankle 5 cm on 200 cm^2 two times daily for 7 days.
  Arms: Diclofenac diethylamine (DDEA) 2.32%/ Placebo gel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of diclofenac diethylamine 2.32 percent (%) gel applied twice daily versus diclofenac diethylamine 1.16% gel applied four times daily for 7 days in participants with acute ankle sprain.

DETAILED DESCRIPTION:
This study is a Phase III, randomized, double blind, multi-center, active controlled, 2-treatment arm, parallel group, non-inferiority study to evaluate the efficacy and safety of diclofenac diethylamine 2.32% gel applied twice daily versus diclofenac diethylamine 1.16% gel applied four times daily for 7 days in participants with acute ankle sprain. The participants who experience an acute Grade I -II ankle sprain within the past 24 hours, and pain on movement of at least 50 millimeter (mm) on a 100 mm visual analogue scale (VAS) and who will meet all inclusion and exclusion criteria will be randomized in a 1:1 ratio, immediately post injury. All participants will receive 4 tubes of study drug, for treatment in morning, noon, late afternoon, and late evening, respectively. The very first dose of study drug will be applied at the study center. The participants will be instructed to apply the gel topically with the finger tips for approximately 1 minute in the morning, at noon, late afternoon, and late evening for 7 days. Each tube will be labeled for use at one of these 4 times. After the randomization visit (Visit 1/baseline visit- Day 1), participants will return to the study site for post baseline visits- Visit 2 (Day 3), Visit 3 (Day 5), and Visit 4 (Day 8 +/- 1 d) to complete efficacy and safety assessments. Baseline safety laboratory test blood samples will be taken at Visit 1. End of study safety laboratory tests will be performed at Visit 4, or in case of early termination on the day of termination. In addition, the participants (ex-clinic) will assess pain intensity and pain relief at frequent intervals on Day 1 and then at each study drug application throughout the rest of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment will be performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant with acute sprain of the lateral ankle on one side only, Grade I-II.
* A participant who had pain-on-movement greater than or equal to (>=) 50 mm on a 100 mm VAS.
* A participant with injury within the past 24 hours before randomization.
* Participant had not taken pain medication within the 24 hours that precedes randomization.Treatment by rest, ice, compression, or elevation (RICE) is authorized prior to randomization. Stable daily doses of acetylsalicylic acid (less than or equal to [<=] 162 mg) taken for at least 30 days prior to the first dose of study medication for non-analgesic reasons may be continued for the duration of the study.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee with no clinically significant/relevant abnormalities in medical history or upon physical examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 14 days after the last dose of assigned treatment.

Exclusion Criteria:

* A participant with Grade I-III sprain of the affected ankle during the past 3 months.
* A participant with Grade II-III sprain, any other significant injury (such as fracture or torn ligament), or surgery (except for skin or nails) of the affected ankle or foot during the past 6 months.
* A participant with pain or instability in the affected ankle attributable to previous ankle sprain or any other trauma.
* A participant with ankle sprain attributable to a known disease affecting the ligaments, such as ligament hyperlaxity due to connective tissue diseases (e.g. Marfan's syndrome, Down's syndrome, Ehlers-Danlos syndrome).
* A participant who has any skin lesion or wound in the area to be treated.
* A participant who intent to undergo surgery during time of participation.
* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant with,in the opinion of the investigator or medically qualified designee, an acute or chronic medical, including other current acute or chronic pain conditions, or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is a pregnant female.
* A participant who is a breastfeeding female.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the Lifestyle Considerations below: a) No special requirement for food and drink prior to safety laboratory evaluations. b) Participants will abstain from caffeine-containing products for 12 hours prior to study visit days (except screening/randomization visit). c) Participants will abstain from strenuous exercise (e.g. heavy lifting, weight training, calisthenics, aerobics) for the duration of the study. Walking at a normal pace will be permitted.
* A participant who has made use of prescription, non-prescription, or dietary supplements, containing NSAIDs, COX-2 inhibitors and other analgesic treatments within 7 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product and during the study.
* A participant with topical analgesics or anti-inflammatory treatment over the previous 30 days in the area to be treated in the study period.
* A participant with evidence of clinically significant laboratory abnormality caused by renal disease (Serum creatinine >=1.5 times the upper limit of normal [ULN]), hepatic disease (ALT or AST >= 2 times the ULN), or subject with allergic disease at screening that may increase the risk associated with study participation.
* A participant with history of regular alcohol consumption exceeding 14 drinks per week (1 drink = 5 ounces [150 milliliter {mL}] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
* A participant who has received treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
* A participant who has previously been enrolled in this study.
* A participant with any physical impairment that would influence the study's efficacy evaluations, in particular POM and the ankle joint function, such as : peripheral or central neurological disease, significant back pain, symptomatic osteoarthritis of the hips, knees or feet, or any painful conditions of the lower extremities (e.g. painful nail, wound, corn, or wart).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (10):
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Chenzhou, Hunan
  - GSK Investigational Site, Dalian, Liaoning
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be grated, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Yin F, Ma J, Xiao H, Ao R, Zhang F, Li W, Wang W, Zeng P, Lu T, Revel FB, Araga M, Patel S, Moreira S, Zhang J, Zhang W. Randomized, double-blind, noninferiority study of diclofenac diethylamine 2.32% gel applied twice daily versus diclofenac diethylamine 1.16% gel applied four times daily in patients with acute ankle sprain. BMC Musculoskelet Disord. 2022 Dec 24;23(1):1125. doi: 10.1186/s12891-022-06077-z. PMID 36566202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 centers in China.
Pre-assignment Details: A total of 313 participants were enrolled into the study and 302 participants were randomized. Of these 150 participants were randomized to Diclofenac diethylamine (DDEA) 2.32 percent (%) gel twice daily (BID) and 152 were randomized to DDEA 1.16% gel four times daily (QID). A total of 288 participants completed the study.
Groups:
- DDEA 2.32% Gel/Placebo: The participants were instructed to apply approximately 2 g DDEA 2.32% gel topically with the fingertips to both sides of affected ankle which corresponds to a region of approximately 200 cm^2 for approximately 1 minute in the morning and in the late afternoon for 7 days. Similarly, participants were instructed to apply placebo gel at noon and in the late evening for 7 days. The very first dose was applied at the study center.
- DDEA 1.16% Gel: The participants were instructed to apply approximately 2 g DDEA 1.16% gel topically with the fingertips to both sides of affected ankle which corresponds to a region of approximately 200 cm^2 for approximately 1 minute in the morning, at noon, in the late afternoon, and in the late evening for 7 days. The very first dose was applied at the study center.
Period: Overall Study
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Started | 150 | 152
Completed | 143 | 145
Not Completed | 7 | 7
Not completed — aspartate aminotransferase (AST) >= 2 times upper limit of normal (ULN) | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Subject did not meet study Criteria | 0 | 1
Not completed — Screened failure, randomized by mistake | 0 | 1
Not completed — Personal reasons | 2 | 4
Not completed — alanine aminotransferase (ALT) >= 2 times ULN | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: Comprise all randomized participants. This population was based on the treatment to which the participant was randomized. Any participant who received a treatment randomization number was considered to have been randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel | Total
Number analyzed (Participants) | 150 | 152 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34 (11.11) | 34.1 (12.41) | 34 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 69 | 133
  Male | 86 | 83 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 152 | 302
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain on Movement (POM) on Day 5 of Treatment as Assessed by a 100 Millimeter (mm) Visual Analogue Scale (VAS)
Description: The investigator performed a movement of the ankle and the pain assessment was done by the participant using a 100 mm VAS by describing ankle pain on movement. The POM was registered by the participant by drawing a perpendicular line on the 100 mm VAS with anchors at 0 = no pain and 100 = extreme pain. Higher scores indicate a worse outcome. Change from Baseline in POM was calculated by subtracting the Baseline value from the Day 5 value.
Time Frame: Baseline and Day 5
Population: Per Protocol (PP) Population: All participants from the Intent-to-Treat (modified) (mITT) population who did not have any major protocol deviations. mITT population comprise all randomized participants who had at least 1 post-Baseline POM VAS assessment.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
mm | -42.36 (1.49) | -43.47 (1.45)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Non-Inferiority — Non-inferiority criteria: if the upper 95% Confidence Interval (CI) of Least Square (LS) mean difference was less than 13 mm then DDEA 2.32% gel BID was concluded as non-inferior; p = 0.5950, ANCOVA; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-3.00 to 5.22], Standard Error of Mean 2.09

2. Secondary Outcome: Number of Participants With Severity of Adverse Events (AEs) Following Dosing With Study Medication
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product or investigational assessment, whether or not considered related to the study product. The investigator or medically qualified designee assessed the intensity for each AE reported during the study and categorized it on the basis of severity as Mild (an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities), Moderate (an event that is sufficiently discomforting to interfere with normal everyday activities or Severe (an event that prevents normal everyday activities).
Time Frame: up to 28 days following last administration of the study product (or last procedure)
Population: Safety Population. It included all participants who were randomized and have received at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 150 | 151
Participants
  Mild | 9 | 8
  Moderate | 2 | 4
  Severe | 0 | 0

3. Secondary Outcome: Change From Baseline of POM on VAS on Day 3 and Day 8 of Treatment Assessed by 100 mm VAS
Description: The investigator performed a movement of the ankle and the pain assessment was done by the participant using a 100 mm VAS by describing ankle pain on movement. The POM was registered by the participant by drawing a perpendicular line on the 100 mm VAS with anchors at 0 = no pain and 100 = extreme pain. Higher scores indicate a worse outcome. Change from Baseline in POM on Day 3 and Day 8 was calculated by subtracting the Baseline value from the Day 3 and Day 8 values respectively.
Time Frame: Baseline and Days 3 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
mm
  Day 3 | -28.29 (1.51) | -25.86 (1.48)
  Day 8: number analyzed (Participants) | 122 | 127
  Day 8 | -55.38 (1.25) | -54.62 (1.23)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.2536, ANCOVA; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-6.61 to 1.75], Standard Error of Mean 2.12 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.6643, ANCOVA; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-4.23 to 2.70], Standard Error of Mean 1.76 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

4. Secondary Outcome: Change From Baseline in Tenderness as Measured by Pressure Algometry on Days 3, 5 and 8
Description: 'Tenderness' was the sensation of pain expressed by a participant when pressure was applied to the body. Tenderness was measured by calibrated algometers in an area of 1 cm^2 at the center of the injured area. The investigator applied the pressure gauge to the marked tender point of maximum sensitivity by placing the gauge at a 90 degree angle vertical to the skin. The participant was instructed to indicate the onset of pain with a verbal cue such as "Yes" or "Stop". Change from Baseline in tenderness on Day 3, 5 and 8 was calculated by subtracting the Baseline value from the Day 3, Day 5 and Day 8 values respectively
Time Frame: Baseline and Days 3, 5 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Newton per square centimeter (N/cm^2)
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
Newton per square centimeter (N/cm^2)
  Day 3 | 6.92 (0.85) | 5.72 (0.83)
  Day 5 | 9.84 (0.97) | 10.76 (0.94)
  Day 8: number analyzed (Participants) | 122 | 127
  Day 8 | 17.06 (1.19) | 15.60 (1.16)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.3118, ANCOVA; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [-1.13 to 3.54], Standard Error of Mean 1.19 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.4937, ANCOVA; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-3.60 to 1.74], Standard Error of Mean 1.35 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5
Statistical Analysis 3: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.3825, ANCOVA; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [-1.83 to 4.74], Standard Error of Mean 1.67 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

5. Secondary Outcome: Changes From Baseline in Difference of Tenderness Between Affected Ankle and Contralateral Ankle Measured by Algometry on Days 3, 5 and 8
Description: 'Tenderness' was the sensation of pain expressed by a participant when pressure was applied to the body. Tenderness was measured by calibrated algometers in an area of 1 cm^2 at the center of the injured area. The investigator applied the pressure gauge to the marked tender point of maximum sensitivity by placing the gauge at a 90 degree angle vertical to the skin. The participant was instructed to indicate the onset of pain with a verbal cue such as "Yes" or "Stop". Difference in tenderness between affected ankle and contralateral ankle is presented. Change from Baseline in tenderness on Day 3, 5 and 8 was calculated by subtracting the Baseline value from the Day 3, Day 5 and Day 8 values respectively.
Time Frame: Baseline and Days 3, 5 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: N/cm^2
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
N/cm^2
  Day 3: number analyzed (Participants) | 122 | 127
  Day 3 | 7.85 (0.90) | 7.59 (0.88)
  Day 5: number analyzed (Participants) | 122 | 127
  Day 5 | 11.34 (0.88) | 12.59 (0.86)
  Day 8: number analyzed (Participants) | 122 | 126
  Day 8 | 16.64 (1.03) | 14.98 (1.01)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.8360, ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-2.23 to 2.75], Standard Error of Mean 1.26 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.3119, ANCOVA; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-3.69 to 1.18], Standard Error of Mean 1.24 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5
Statistical Analysis 3: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.2535, ANCOVA; Mean Difference (Final Values) = 1.66, 95% CI 2-sided [-1.20 to 4.52], Standard Error of Mean 1.45 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

6. Secondary Outcome: Change From Baseline in Ankle Joint Function (Karlsson Scoring Scale) on Days 3, 5 and 8
Description: Ankle Joint Function was assessed by the participants using Karlsson Scoring Scale. The scoring scale measured recovery of ankle joint function after an acute ligament injury. Assessments were made in the following eight categories (score): pain (20), swelling (10), instability (subjective) (15), stiffness (5), stair climbing (10), running (10), work activities (15), and the use of a support device (5). The total score ranges in value from 0 (worst possible score) to 90 (best possible score). Change from Baseline in the ankle joint function on Days 3, 5 and 8 was calculated by subtracting the Baseline value from the Day 3, Day 5 and Day 8 values respectively.
Time Frame: Baseline and Days 3, 5 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
Scores on a scale
  Day 3 | 16.26 (1.07) | 15.52 (1.05)
  Day 5 | 27.94 (1.46) | 28.22 (1.43)
  Day 8: number analyzed (Participants) | 122 | 127
  Day 8 | 41.87 (1.59) | 39.75 (1.56)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.6242, ANCOVA; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-2.23 to 3.71], Standard Error of Mean 1.51 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.8905, ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-4.33 to 3.77], Standard Error of Mean 2.06 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5
Statistical Analysis 3: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.3439, ANCOVA; Mean Difference (Final Values) = 2.12, 95% CI 2-sided [-2.29 to 6.54], Standard Error of Mean 2.24 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

7. Secondary Outcome: Change From Baseline in Circumference of Affected Ankle (Swelling) as Measured by Figure of Eight Method on Days 3, 5 and 8
Description: Each participant was seated comfortably in a long sitting position with both feet extended beyond the end of the plinth in a slight dorsiflexion position. The Figure of Eight Method was applied to both feet and the tape measure was wrapped around the ankle along the following course: the beginning of the tape was placed midway between the tibialis anterior tendon and lateral malleolus and was then continued across anatomically defined points in the form of a figure of eight around the ankle joint. The tape localization of the first measurement was marked with an appropriate marker. Each ankle was measured three times and the average was calculated. Change from Baseline in circumference on Days 3, 5 and 8 was calculated by subtracting the Baseline value from the Day 3, Day 5 and Day 8 values respectively.
Time Frame: Baseline and Days 3, 5 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Centimeter (cm)
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
Centimeter (cm)
  Day 3: number analyzed (Participants) | 122 | 127
  Day 3 | -0.42 (0.09) | -0.24 (0.09)
  Day 5: number analyzed (Participants) | 122 | 127
  Day 5 | -0.97 (0.10) | -0.57 (0.10)
  Day 8: number analyzed (Participants) | 122 | 126
  Day 8 | -1.25 (0.10) | -0.87 (0.10)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.1554, ANCOVA; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.44 to 0.07], Standard Error of Mean 0.13 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.0047, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.66 to -0.12], Standard Error of Mean 0.14 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5
Statistical Analysis 3: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.0082, ANCOVA; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.66 to -0.10], Standard Error of Mean 0.14 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

8. Secondary Outcome: Change From Baseline in Difference of Circumference (Swelling) Between Affected Ankle and Contralateral Ankle by Figure of Eight Method on Days 3, 5 and 8
Description: Each participant was seated comfortably in a long sitting position with both feet extended beyond the end of the plinth in a slight dorsiflexion position. The Figure of Eight Method was applied to both feet and the tape measure was wrapped around the ankle along the following course: the beginning of the tape was placed midway between the tibialis anterior tendon and lateral malleolus and was then continued across anatomically defined points in the form of a figure of eight around the ankle joint. The tape localization of the first measurement was marked with an appropriate marker. Each ankle was measured three times and the average was calculated. Difference of circumference (swelling) between affected ankle and contralateral ankle is presented. Change from Baseline in circumference on Days 3, 5 and 8 was calculated by subtracting the Baseline value from the Day 3, Day 5 and Day 8 values respectively.
Time Frame: Baseline and Days 3, 5 and 8
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 128
cm
  Day 3: number analyzed (Participants) | 122 | 127
  Day 3 | -0.41 (0.07) | -0.29 (0.06)
  Day 5: number analyzed (Participants) | 122 | 127
  Day 5 | -0.83 (0.07) | -0.66 (0.06)
  Day 8: number analyzed (Participants) | 122 | 126
  Day 8 | -1.12 (0.06) | -0.92 (0.06)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.2182, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.30 to 0.07], Standard Error of Mean 0.09 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 3
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.0574, ANCOVA; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.36 to 0.01], Standard Error of Mean 0.09 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5
Statistical Analysis 3: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.0194, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.37 to -0.03], Standard Error of Mean 0.08 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 8

9. Secondary Outcome: Sum of Pain Intensity Difference (SPID) From 0 to 24 Hours Post First Dose (Day 1) and From 96 to 120 Hours Post First Dose (Day 5)
Description: Pain intensity was assessed in the diary on a categorical scale ranging from 0 to 3, where 0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain. A higher value indicates more severe pain. Pain intensity was assessed at Baseline (immediately prior to first dose) and every 2 hours (after starting study product) until the participant went to bed on the evening of Day 1. The same assessment and recording frequency were also followed starting with the first dose on Day 5.
Time Frame: 0 to 24 hours (Day 1) and 96 to 120 hours (Day 5) post first dose
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 126
Scores on a scale
  Sum of 0 - 12 hours post first dose (Day 1) | 15.80 (0.583) | 15.43 (0.574)
  Sum of 96 - 120 hours post first dose (Day 5) | 9.80 (0.512) | 10.29 (0.503)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.6545, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-1.250 to 1.986], Standard Error of Mean 0.821 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 1
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.4924, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.915 to 0.924], Standard Error of Mean 0.721 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5

10. Secondary Outcome: Total Pain Relief (TOTPAR) From 0 to 24 Hours Post First Dose (Day 1) and From 96 to 120 Hours Post First Dose (Day 5)
Description: Pain relief was assessed in the diary on a categorical scale ranging from 0 to 4, where 0 = no relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief. A higher value indicates greater pain relief. Pain relief was assessed at Baseline (immediately prior to first dose) and every 2 hours (after starting study product) until the participant went to bed on the evening of Day 1. The same assessment and recording frequency were also followed starting with the first dose on Day 5.
Time Frame: 0 to 24 hours (Day 1) and 96 to 120 hours (Day 5) post first dose
Population: PP Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 122 | 126
Scores on a scale
  Sum of 0-12 hours post first dose (Day 1) | 8.47 (0.585) | 8.53 (0.575)
  Sum of 96-120 hours post first dose (Day 5) | 28.48 (1.030) | 27.68 (1.014)
Statistical Analysis 1: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.9491, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.675 to 1.570], Standard Error of Mean 0.823 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 1
Statistical Analysis 2: Comparison: DDEA 2.32% Gel/Placebo vs DDEA 1.16% Gel; Test type: Other; p = 0.5820, ANCOVA; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-2.059 to 3.659], Standard Error of Mean 1.451 — DDEA 2.32% gel vs DDEA 1.16% gel, Day 5

11. Secondary Outcome: Mean Number of Rescue Medication Tablets Used to Treat Ankle Pain
Description: Participants were instructed to take only the rescue medication provided for pain in the ankle or any other pain (for example, headache) or fever (for example, due to common cold) they experienced during the trial. One tablet was taken, repeated after at least 4 hours, if needed, up to a maximum of 2000 milligram (mg) (4 tablets) per day. No rescue medication was allowed within 6 hours prior to the study visits or within 12 hours of study Visit 3.
Time Frame: Up to Day 8
Population: ITT Population. Only those participants who used rescue medication were analyzed.
Measure: Mean (Standard Deviation); unit: Number of Tablets
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 8 | 12
Number of Tablets | 2.4 (2.39) | 2.6 (2.19)

12. Secondary Outcome: Number of Days on Which Rescue Medication Was Used to Treat Ankle Pain
Description: Data was not estimable as end date data for rescue medication use was not collected.
Time Frame: Up to Day 8
Population: ITT Population. Data was not collected for this outcome measure.
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to 28 days following last administration of the study product (or last procedure).
Description: Treatment emergent AEs were defined as any new AE that occurred on or after the date/time of the first administration of study product, or any pre-existing AE that was considered to have worsened on or after the date/time of the first administration of study product.
Arm/Group | DDEA 2.32% Gel/Placebo | DDEA 1.16% Gel
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/151
Other Adverse Events (participants affected / at risk) | 11/150 | 12/151
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DDEA 2.32% Gel/Placebo (N=150) | DDEA 1.16% Gel (N=151)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Application site inflammation (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Endometrial thickening (Reproductive system and breast disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04052620/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT04052620/SAP_001.pdf